CLINICAL TRIAL: NCT03146455
Title: Establishment for Thromboelastography Normal Reference Values of Healthy Adults in China Hunan Province: A Multicenter Observational Study
Brief Title: Thromboelastography Normal Reference Values in China Hunan Province
Status: Completed | Type: Observational
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Collaborators: Second Xiangya Hospital of Central South University (Other); Hunan Provincial People's Hospital (Other); Hunan Cancer Hospital (Other); Changsha Central Hospital (Other)
Responsible Party: Principal Investigator, xy3transfusion, Director, Blood transfusion, The Third Xiangya Hospital of Central South University
Other Study IDs: ThirdXiangyaHCSU
Record Dates: First submitted 2017-05-07; First posted 2017-05-10 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Coagulopathy; Blood Transfusion Complication
Keywords: Thrombelastograghy; reference ranges; racial; geographic; Blood Transfusion
MeSH Terms: conditions — Hemostatic Disorders; Transfusion Reaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health adults: (1) 18< Age <65, and Han Chinese residents living in Hunan more than 3 years. (2) Health examination population who physical examination, assistant examination and serological examination were normal; Not suffer from other diseases last 3 months; Not take any medication last 7 days.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The purpose of this study was to establish the normal reference range of Thrombelastogram parameters in Hunan by a multicenter study, and to analyze the specificity of Thrombelastogram detection and the influence of gender, age and blood type on Thrombelastogram. The study will provide basic data and statistical basis for the establishment of normal reference range of Thrombelastogram in Hunan.

DETAILED DESCRIPTION:
Thrombelastograghy (TEG) is an important test to assess the blood coagulation function to monitor the whole process of perioperative coagulation. TEG can evaluate the coagulation cascade, from platelet aggregation, clot strengthening and fibrin cross-linking to eventually clot lysis in small volume of whole blood. The reference range is one important element to influence the TEG results. At present, a number of studies have shown that reference range of TEG exists significant differences between different racial and geographic. At the same time, reagent manufacturers also suggested that each TEG laboratory should establish its own reference range. So it is important to establish our own reference range of TEG to guide the clinical blood transfusion and treatment.

ELIGIBILITY:
Inclusion Criteria:

(1) 18< Age <65, and Han Chinese residents living in Hunan more than 3 years. (2) Health examination population who physical examination, assistant examination and serological examination were normal; Not suffer from other diseases last 3 months; Not take any medication last 7 days.

Exclusion Criteria:

1. Informed refusal. 2. Pregnancy, woman with menstrual period; volunteers who suffer from hematological system diseases such as hemorrhagic or thrombotic disease and take medicines that affect the function of blood coagulation (clopidogrel and aspirin, warfarin, rivaroxaban, dipyridamole, oral contraceptives, estrogen, antibiotics and traditional Chinese medicine related with blood coagulation, etc.) 3. Volunteers who have a history of liver disease, immune system disease, allergy and other disease within the last 3 months were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Permanent resident in Hunan, 18< Age <65.
Sampling Method: Probability Sample
Enrollment: 498 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-03-10 (Actual)

PRIMARY OUTCOMES:
thromboelastography normal reference values | 2017.6.1-2017.12.1
  The subjects with normal routine coagulation test results would be included.Thromboelastography was performed by using TEG-5000 TEG-CK (Hemostasis System, USA), and the parameters were recorded. Parameters includes R (coagulation reaction time, initial fibrin formation time), K (Coagulation time), α (α-angle, thrombosis rate), MA (maximum amplitude, absolute agglutination strength of reactive blood clot), LY30 (fibrinolysis rate with 30 min after MA determination) and CI (integrated coagulation index).

CONTACTS AND LOCATIONS:
Locations (1):
- Third Xingya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pfanner G, Koscielny J, Pernerstorfer T, Gutl M, Perger P, Fries D, Hofmann N, Innerhofer P, Kneifl W, Neuner L, Schochl H, Kozek-Langenecker SA; Austrian Society for Anaesthesia, Resuscitation and Intensive Care. [Preoperative evaluation of the bleeding history. Recommendations of the working group on perioperative coagulation of the Austrian Society for Anaesthesia, Resuscitation and Intensive Care]. Anaesthesist. 2007 Jun;56(6):604-11. doi: 10.1007/s00101-007-1182-0. German. PMID 17522829
- [Background] Sun W, Jeleniowski K, Zhao X, Shen P, Li D, Hammond JA. Thromboelastography (TEG)-based algorithm reduces blood product utilization in patients undergoing VAD implant. J Card Surg. 2014 Mar;29(2):238-43. doi: 10.1111/jocs.12302. PMID 24734284
- [Background] Wesley MC, McGowan FX, Castro RA, Dissanayake S, Zurakowski D, Dinardo JA. The effect of milrinone on platelet activation as determined by TEG platelet mapping. Anesth Analg. 2009 May;108(5):1425-9. doi: 10.1213/ane.0b013e3181981fbe. PMID 19372315
- [Background] Wang SC, Shieh JF, Chang KY, Chu YC, Liu CS, Loong CC, Chan KH, Mandell S, Tsou MY. Thromboelastography-guided transfusion decreases intraoperative blood transfusion during orthotopic liver transplantation: randomized clinical trial. Transplant Proc. 2010 Sep;42(7):2590-3. doi: 10.1016/j.transproceed.2010.05.144. PMID 20832550
- [Background] Ak K, Isbir CS, Tetik S, Atalan N, Tekeli A, Aljodi M, Civelek A, Arsan S. Thromboelastography-based transfusion algorithm reduces blood product use after elective CABG: a prospective randomized study. J Card Surg. 2009 Jul-Aug;24(4):404-10. doi: 10.1111/j.1540-8191.2009.00840.x. PMID 19583608
- [Background] Zambruni A, Thalheimer U, Leandro G, Perry D, Burroughs AK. Thromboelastography with citrated blood: comparability with native blood, stability of citrate storage and effect of repeated sampling. Blood Coagul Fibrinolysis. 2004 Jan;15(1):103-7. doi: 10.1097/00001721-200401000-00017. PMID 15166952
- [Background] Subramanian A, Albert V, Saxena R, Agrawal D, Pandey RM. Establishing a normal reference range for thromboelastography in North Indian healthy volunteers. Indian J Pathol Microbiol. 2014 Jan-Mar;57(1):43-50. doi: 10.4103/0377-4929.130896. PMID 24739830
- [Background] Ji HW, Ma L, Gao XR, Liu N, Zhang Y, Wang Y, Ma ZX, Wang Y, Wang J, Fu X, Xiong Q, Qi HM. [Establishment of normal reference values for thromboelastography on Chinese population in Beijing]. Zhonghua Yi Xue Za Zhi. 2011 Apr 12;91(14):980-3. Chinese. PMID 21609551